CLINICAL TRIAL: NCT06665841
Title: Correlation Between Selenium Levels in Human Tissues and HPV-related Cervical Lesions and Outcomes
Acronym: SeHPV
Status: Not yet recruiting | Type: Observational
Sponsor: Second Affiliated Hospital of Wenzhou Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: SAHoWMU-CR2024-07-220
Record Dates: First submitted 2024-10-28; First posted 2024-10-30 (Actual); Last update posted 2024-10-30 (Actual); Status verified 2024-10

CONDITIONS: Cervical Intraepithelial Neoplasia (CIN); Cervical Cancer; Persistent HPV Infection
Keywords: Selenium; Persistent HPV Infection; Cervical Lesions
MeSH Terms: conditions — Uterine Cervical Dysplasia; Uterine Cervical Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Trial volunteers: Trial volunteers refer to healthy individuals undergoing physical examinations at our hospital or recruited healthy university students.
- Cervical lesions: Patients with cervical lesions, including those with uterine fibroids, cervical cancer, endometrial cancer, and ovarian cancer.
- persistent HPV infection: Persistent HPV infection refers to the infection by the same type of HPV for more than 12 months.
- Non-persistent HPV infection: Non-persistent HPV infection refers to the absence of HPV infection.

SUMMARY:
This study investigates the relationship between selenium levels in human tissues and the persistence of HPV (human papillomavirus) infection, particularly focusing on cervical-related lesions. The main objectives are to explore the correlation between selenium levels in different body samples (hair, nails, urine, and blood) and to evaluate selenium's potential protective effects against HPV persistence and its progression to cervical lesions.

Key goals of the study include:

Determining whether non-invasive monitoring (e.g., hair, nails, urine) can accurately reflect blood selenium levels.

Understanding how selenium levels fluctuate in women with persistent HPV infection, and whether selenium supplementation can reduce the risk of HPV-related cervical disease progression.

Exploring selenium's role in enhancing immune function, especially in older adults, to help clear HPV infection.

By recruiting volunteers for selenium level testing and tracking HPV-positive women over time, this research aims to provide evidence on the effectiveness of selenium in preventing cervical cancer progression and potentially clearing HPV infections.

DETAILED DESCRIPTION:
This prospective study aims to explore the impact of selenium levels in human tissues on the progression of HPV-related cervical lesions and to identify the most appropriate biological samples for monitoring selenium levels. The research is divided into three parts:

Part 1: Volunteer Recruitment and Selenium Level Assessment Healthy volunteers, such as those undergoing regular medical check-ups or university students, will be recruited. Selenium levels in various biological samples-blood, hair (scalp or pubic), urine, and nails-will be measured. The primary goal is to assess the correlation between selenium levels in these different tissues to determine whether non-invasive samples (hair, nails, urine) could be used as reliable indicators of blood selenium levels.

Part 2: Patient Group Sample Collection Samples will be collected from hospitalized patients diagnosed with conditions such as uterine fibroids, cervical cancer, endometrial cancer, and ovarian cancer. These samples will include blood, hair (scalp or pubic), urine, and nails, with the same goal of determining the correlation between selenium levels in various tissues. This part of the study will help assess selenium levels in patients with reproductive system diseases and evaluate any differences compared to healthy individuals.

Part 3: HPV Persistent Infection Group Women with persistent HPV infection (defined as infection with the same HPV type for more than 12 months) will be selected from the gynecology clinic, along with a control group of women with non-persistent HPV infection. Selenium levels and immune function will be evaluated at baseline and again after 12 months. Comparisons will be made between the two groups to assess changes in selenium levels and immune function. Additionally, patients with HPV-related cervical lesions (e.g., CIN or cervical cancer) and those with normal cervical tissues will have their serum selenium levels and immune function assessed.

This part of the study will also include the collection of blood, hair (scalp or pubic), urine, and nail samples from HPV-persistent patients. These patients will be divided into three groups: (1) no treatment, (2) interferon treatment (standard clinical practice), and (3) interferon combined with selenium supplementation. The patients will be monitored for 6 and 12 months to observe changes in HPV status (whether the infection clears or persists) and to analyze selenium levels, immune function, and disease progression in CIN I patients.

Selenium supplementation, provided in the form of nano-selenium capsules, will be administered based on the selenium status determined from the external lab results. Patients will be divided into three groups based on their selenium levels:

Normal selenium levels: 50 µg selenium supplement, taken twice daily. Selenium deficiency: 100 µg selenium supplement, taken twice daily. Severe selenium deficiency: 150 µg selenium supplement, taken twice daily. The study will employ various statistical methods, including correlation analysis, univariate and multivariate analysis, and variance analysis, to evaluate the results. The findings will help determine whether selenium supplementation can aid in HPV clearance, slow the progression of cervical lesions, and enhance immune function, particularly in selenium-deficient individuals.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 to 65 years;
* No history of sexual activity within the past 3 days;
* No history of cervical surgery;
* No history of using contraceptives, hormone therapy, or exposure to metals;
* No history of cardiovascular, cerebrovascular, liver, kidney, or thyroid diseases;
* All participants must sign a written informed consent form prior to sampling and agree to cooperate with the study.

Exclusion Criteria:

* Previous diagnosis of HPV positivity and those who have received treatment;
* Pregnant individuals;
* Individuals who refuse to cooperate.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — This study is open to individuals who self-identify as female or any gender identity that aligns with the biological sex of female, including transgender women and non-binary individuals who consider themselves female.
Study Population: Part 1 of the Study: Study Subjects: Volunteers (individuals undergoing routine health examinations or university students) Part 2 of the Study: Study Subjects: Hospitalized patients (e.g., vaginal uterine prolapse, uterine fibroids, cervical cancer, endometrial cancer, ovarian cancer, etc.) Part 3 of the Study: Study Subjects: First-time HPV infection patients from the gynecology outpatient clinic of our hospital.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2024-11-01 (Estimated); Primary Completion 2027-06-30 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Selenium Level Assessment: | At enrollment, 6 months after enrollment, and 12 months after enrollment
  Measurement of serum selenium content: Determined by atomic fluorescence spectrometry / inductively coupled plasma mass spectrometry.

SECONDARY OUTCOMES:
Immune Function Evaluation | At enrollment, 6 months after enrollment, and 12 months after enrollment
  Complete blood count: White blood cell count, neutrophils, lymphocytes, monocytes, red blood cells, hemoglobin, platelets, CRP. Analysis of immune cells in peripheral blood (flow cytometry): B cells; T cells; NK cells; monocytes.
HPV and TCT Detection, and Definition of HPV Clearance | At enrollment, 6 months after enrollment, and 12 months after enrollment
  HPV detection: Real-time quantitative PCR; TCT detection: Cervical cells are assessed using a liquid-based thin-layer cytology system and classified cytologically.
  Definition of HPV clearance:
  * Ineffective: HPV subtype remains positive or increases other subtypes; ② Improvement: ≥1 HPV positive subtype becomes negative while still having HPV infection; ③ Complete clearance: All HPV subtypes become negative.

IPD SHARING:
Plan to Share IPD: No
The study will be used for publication in academic journals, and therefore individual participant data (IPD) will not be shared.